CLINICAL TRIAL: NCT01231750
Title: A Randomized, Placebo-Controlled, Cross-Over Study to Assess the Safety and Efficacy of TOPical CAPsaicin With Stable Angina (TOPCAP)
Brief Title: Efficacy of Topical Capsaicin Cream for Stable Angina
Acronym: TOPCAP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to identify study population to achieve number expected
Sponsor: Neal Weintraub (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor-Investigator, Neal Weintraub, Professor, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UC 060559
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Results first posted 2015-06-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Stable Angina
MeSH Terms: conditions — Angina, Stable | interventions — Capsaicin; Drugs, Generic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.1% Capsaicin Cream (Active Comparator): 0.1% capsaicin cream spread 8cm x 15cm on abdomen, once, 45 minutes prior to exercise
  Interventions: Drug: Capsaicin
- Placebo Cream (Placebo Comparator): Inactive cream, 4cm spread 8cm x 15cm on the abdomen, once, 45 minutes prior to exercise
  Interventions: Other: Placebo cream

INTERVENTIONS:
Drug: Capsaicin — 0.1% topical cream,4cm spread over 8cm x 15cm area on skin, one time, 45 minutes prior to exercise
  Other Names: capsaicin cream 0.1%, generic
  Arms: 0.1% Capsaicin Cream
Other: Placebo cream — cream, 4cm spread over 8cm x 15cm area of skin
  Other Names: cream, placebo
  Arms: Placebo Cream

SUMMARY:
The purpose of this study is to test the hypothesis that application of topical capsaicin in patients with stable angina will result in improved exercise tolerance and reduced cardiac ischemia.

DETAILED DESCRIPTION:
Patients with stable angina on medical therapy who are capable of exercising on a treadmill and have an interpretable ECG for ischemia will be enrolled in the study, which entails performing two treadmill tests approximately one week apart following topical treatment with placebo cream or topical capsaicin (randomized in crossover fashion). Patients will be monitored for exercise tolerance, anginal symptoms, ECG for ischemia/arrhythmia, and hemodynamic responses.

ELIGIBILITY:
Inclusion Criteria:

* > or = 3 month history of chronic, stable, angina triggered by physical effort or mental/emotional stress
* documented stress-induced ST depression, reversible perfusion imaging, or wall motion abnormality or CAD >50%
* Canadian Cardiovascular (CV) Class I-III
* Receiving medical therapy for > or = 2 months
* Ability to perform Bruce Protocol treadmill test
* non-pregnant female

Exclusion Criteria:

* unstable angina
* revasc within 2 months
* Myocardial infarction (MI) within 2 months
* congestive heart failure (CHF) hospitalization within 2 months
* New York Heart Association (NYHA) class III or IV
* left ventricular ejection fraction (LVEF) < 25%
* abnormal ECG; Acute changes on ECG
* Currently receiving treatment with investigational drugs/devices
* Uncontrolled hypertension
* contraindication to exercise stress testing
* allergy to red peppers or capsaicin
* skin deformity, scar, or rash at application site
* abdominal surgery within 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faisal M Khan, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Physicians, Inc, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment goal not met.
Pre-assignment Details: Inclusion and exclusion criteria proved a large screening volume to yield few participants.
Groups:
- 0.1% Capsaicin Cream First, Then Placebo: Capsaicin : 0.1% topical cream,4cm spread over 8cm x 15cm area on skin, one time, 45 minutes prior to exercise
- Placebo First, Then 0.1% Capsaicin: Inactive substance, 4cm spread 8cm x 15cm on skin, once, 45 minutes prior to exercise
  Placebo cream : cream, 4cm spread over 8cm x 15cm area of skin
Period: Overall Study
Arm/Group | 0.1% Capsaicin Cream First, Then Placebo | Placebo First, Then 0.1% Capsaicin
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.1% Capsaicin Cream First, Then Placebo | Placebo First, Then 0.1% Capsaicin | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Symptom-limited Exercise Duration as an Indicator of Exercise Capacity
Description: Subjects walked on the treadmill as long as they could tolerate, symptom-limited.
Time Frame: Application was 45 minutes prior to exercise
Population: Data collected are no longer accessible.
Arm/Group | 0.1% Capsaicin Cream First, Then Placebo | Placebo First, Then 0.1% Capsaicin
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Time-to-onset of 1mm ST Segment Depression
Description: Continuous ECG was recorded during exercise. ECG was reviewed by a board-certified cardiologist.
Time Frame: Application was 45 minutes prior to exercise
Population: Data collected are no longer accessible.
Arm/Group | 0.1% Capsaicin Cream First, Then Placebo | Placebo First, Then 0.1% Capsaicin
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Time-to-onset of Angina or Angina Equivalent Symptoms
Description: Onset of angina or angina-equivalent symptoms was assessed from beginning of exercise.
Time Frame: Application was 45 minutes prior to exercise
Population: Data collected are no longer accessible.
Arm/Group | 0.1% Capsaicin Cream First, Then Placebo | Placebo First, Then 0.1% Capsaicin
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Maximal ST Depression
Description: Exercise ECG data was reviewed by a board certified cardiologist to assess maximal ST depression.
Time Frame: Application was 45 minutes prior to exercise
Population: Data collected are no longer accessible.
Arm/Group | 0.1% Capsaicin Cream First, Then Placebo | Placebo First, Then 0.1% Capsaicin
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Maximal Estimated Workload (in METS)
Description: Maximal estimated workload (in METS) was measured during exercise tolerance test (ETT).
Time Frame: Application was 45 minutes prior to exercise
Population: Data collected are no longer accessible.
Arm/Group | 0.1% Capsaicin Cream First, Then Placebo | Placebo First, Then 0.1% Capsaicin
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Magnitude of Reversible Perfusion Defect in SPECT With Wall Motion Assessment (Phase 2)
Description: Phase 2 of the study involving nuclear imaging was not done because the study was stopped early for lack of enrollment.
Time Frame: Phase 2 was not done.
Arm/Group | 0.1% Capsaicin Cream First, Then Placebo | Placebo First, Then 0.1% Capsaicin
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Severity of Angina Was Measured.
Description: Severity of angina was measured using numerical score 1 to 10, where 10 is the worst intensity and 1 is the least.
Time Frame: Application was 45 minutes prior to exercise
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 18 months
Description: Adverse events were assessed, but none observed.
Arm/Group | 0.1% Capsaicin Cream First, Then Placebo | Placebo First, Then 0.1% Capsaicin
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes